CLINICAL TRIAL: NCT06085742
Title: BRE-08: A Phase II Study of an All-Oral Adjuvant Chemotherapy Regimen of Cyclophosphamide, Methotrexate, and Capecitabine (CMC) for Early-Stage Breast Cancer
Brief Title: BRE-08 Phase II Study of CMC Regimen for Early Stage Breast Cancer
Acronym: BRE-08
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Abiola Ibraheem, Principal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0429
Record Dates: First submitted 2023-10-09; First posted 2023-10-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Methotrexate; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CMC orally (Other): All agents in CMC are oral and conform to a 3-week = 1 cycle regimen. All subjects will receive Cyclophosphamide 60mg/m2 PO once a day (21 continuous days) Methotrexate 10mg/m2 PO BID on days 1, 8, and 15 Capecitabine 825mg/m2 PO BID on days 1-14
  Interventions: Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Capecitabine

INTERVENTIONS:
Drug: Cyclophosphamide — 60mg/m2 PO once a day (21 continuous days)
Drug: Methotrexate — 10mg/m2 PO BID on days 1, 8, and 15
Drug: Capecitabine — 825mg/m2 PO BID on days 1-14

SUMMARY:
This is a non-randomized, single arm phase 2 trial of oral CMC based on conversion of doses that would be delivered with conventional metronomic CMF chemotherapy.

DETAILED DESCRIPTION:
Participants who require adjuvant radiotherapy for locoregional management may opt to initiate radiotherapy following the fourth cycle of CMC with the final 4 cycles held during radiotherapy. Following completion of radiation therapy, participants may then resume with cycle 5 of CMC. The washout period before and after radiation therapy is a minimum of 2 weeks. Alternatively, patients may receive adjuvant radiotherapy after the completion of the final (8) cycle of CMC.

The study team will collect data on cyclophosphamide, methotrexate, and capecitabine compliance at routine clinical visits every 3 weeks. In addition, standard electrolyte, chemistry and liver function laboratory monitoring will be conducted at each clinic visit

ELIGIBILITY:
Inclusion Criteria:

I• Age ≥ 18 years of age at time of consent

* ECOG performance status 0, 1, or 2
* Histologically confirmed invasive breast cancer documented by biopsy or surgical excision.
* Underwent potentially curative resection of primary breast tumor(s) with no gross residual local-regional disease (patients with microscopically positive margins are eligible if adjuvant radiotherapy is planned), with most recent breast or axillary surgery < 90 days prior to date of signed consent.
* No evidence of distant metastatic disease
* No prior systemic therapy for this cancer other than pre-operative endocrine therapy
* Treating Oncologist recommends adjuvant chemotherapy without concurrent biologic/targeted therapy. Patients may receive a CDK4/6 inhibitor after completion of all study treatment, concurrently with adjuvant endocrine therapy. Patients with a germline pathogenic/likely pathogenic variant in a DNA homologous repair gene (e.g. BRCA1, BRCA2, PALB2) may receive adjuvant PARP inhibitor therapy after completion of all study treatment.
* Tumor is estrogen receptor (ER)-positive (> 10% by IHC) and/or progesterone receptor (PR)-positive (> 10% by IHC), HER2-negative by IHC or FISH according to 2018 ASCO-CAP guidelines.
* AJCC pathologic stage:

  o pT1-3/pN0-2 based on sentinel lymph node biopsy or axillary dissection
* High risk gene expression profile (either luminal B on MammaPrint/BluePrint, or Recurrence Score > 25 on Oncotype Dx). Study participants are not required to have a high-risk gene expression profile if they have a clinical high-risk tumor, defined as:

Age < 50 and any of the following:

* Involvement of 1-3 axillary lymph nodes with metastatic carcinoma (pN1mic/N1)
* grade 1 tumor > 3 cm; or grade 2 tumor > 2 cm; or grade 3 tumors > 1 cm (size based on pathological assessment of the maximal dimension of the invasive component of the tumor)
* pT1c-T2 and Ki-67 > 20%
* Presence of lymphovascular invasion stage IIIA (pT3/pN1 or pT1-3/pN2)

Age > 50 and any of the following:

* Primary tumor > 5 cm (pT3)
* stage IIIA (pT3/pN1 or pT1-3/pN2)

  * Adequate organ function as defined in Table 1. All screening labs to be obtained within 30 days prior to registration.
  * Patients with synchronous bilateral primary breast tumors or multiple ipsilateral primary breast tumors are eligible if the treating Oncologist determines that the CMC regimen is appropriate therapy for all primary tumors requiring chemotherapy.
  * Able to provide written informed consent and HIPAA authorization for release of personal health information.
  * Women of childbearing potential must agree to use 2 methods of birth control, at least one being a barrier form of contraception if they are sexually active with a male partner unless they are considered highly unlikely to conceive as defined in section 8.6, and cannot be pregnant or breast-feeding. A negative serum or urine pregnancy test is required per institutional practice guidelines.
  * As determined at the discretion of the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.
  * Patients with history of HIV/AIDS (acquired immunodeficiency syndrome) are eligible for this study if they are receiving anti-retroviral therapy and it does not include any medications known to alter metabolism or tolerability of component drugs in the CMC regimen (see Appendix), and either of the following criteria are met:

    * Patients without a history of AIDS-defining opportunistic infections.
    * Patients with a history of AIDS-defining opportunistic infections, but they have not had an opportunistic infection within the past 12 months.
  * Patients with Hepatitis B (HBV): chronic carriers of HBV infection (HBsAg-positive) or individuals who have serologic evidence of a resolved prior HBV infection (i.e., HBsAg-negative and anti-HBc-positive) are eligible if they are receiving appropriate suppressive antiviral therapy that does not include medications known to alter metabolism or tolerability of component drugs in CMC (see Appendix) prior to initiation of cancer therapy, and liver function tests meet study eligibility criteria.
  * Patients with Hepatitis C (HCV): patients with a history of HCV infection who have completed curative antiviral treatment are eligible if the HCV RNA viral load is below the limit of quantification within 90 days of study enrollment. Patients on concurrent HCV treatment must have HCV RNA viral load below the limit of quantification within 30 days of study enrollment. Patients must also meet liver function test eligibility requirements and antiviral therapy does not include medications known to alter metabolism or tolerability of component drugs in CMC.

Exclusion Criteria

Subjects meeting any of the criteria below are ineligible for this study:

* Prior cytotoxic chemotherapy for this breast cancer
* Any investigational agents administered during or within 2 weeks prior to start of CMC chemotherapy
* AJCC stage IIIB-IIIC or stage IV
* Active infection requiring systemic therapy
* Untreated HIV/AIDS
* Documented DYPD deficiency
* Pregnant or nursing
* Require anticoagulation with warfarin. Anticoagulation with low molecular weight heparins, heparin, or direct oral anticoagulants (DOACs) is permitted.
* Any prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of this investigational regimen, as determined by the treating medical oncologist.
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial.
* Other major comorbidity (e.g. advanced cardiopulmonary disease, uncontrolled diabetes mellitus) that may affect the safety or efficacy assessment of this investigational regimen, as determined by study PI
* Inability to swallow pills
* Any medical condition interfering with absorption of oral medications
* Any contraindication for any chemotherapy drug used in the CMC regimen
* Active and ongoing use of medicines known to alter metabolism or tolerability of component drugs in CMC.
* Prisoners
* Unable or unwilling to take a large number of oral pills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2034-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
Relative Dose Intensity (RDI) in patients treated with the CMC regimen. RDI is defined as the sum total of delivered drug in mg/m2/week for each drug in the CMC regimen per the number of participants that have equal to or greater than 85% | 1 year
  Number of participants that have RDI of the CMC regimen is equal to or greater than 85%

SECONDARY OUTCOMES:
Safety of oral CMC regime per the number of participants experiencing adverse events | 1 year
  Number of participants having adverse event using the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5
Invasive Disease Free Survival (iDFS) | 10 years
  Number of participants that have iDFS, defined as the time from enrollment to
  documentation of the first of the following: invasive cancer in the ipsilateral breast/chest wall or regional nodes, contralateral invasive breast or regional nodes, distant metastases, or death from any cause
Distant Disease Free Survival (DDFS) | 10 years
  Number of participants that have DDFS defined as the time from enrollment to documentation of distant metastases or death from any cause.
Overall Survival (OS) | 10 years
  Number of participants that have OS defined as the time from study enrollment to the date of the subject's death
Participant outcomes using the Quality of Life (QOL) and EORTC QOL-C30 questionnaires | 10 years
  Number of participants having good outcome versus low outcomes. High score means worse health outcomes and low score means better health outcomes
Protocol therapy interruption | 10 years
  Number of participants that have protocol therapy interruption
Discontinuation of protocol therapy | 10 years
  Number of participants that have discontinuation of protocol therapy
Rates of dose reduction of cyclophosphamide | 10 years
  Number of participants that have dose reduction of cyclophosphamide
Rates of dose reduction of methotrexate | 10 years
  Number of participants that have dose reduction of methotrexate
Rates of dose reduction of capecitabine | 10 years
  Number of participants that have dose reduction of capecitabine

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois, Chicago, Illinois, United States